CLINICAL TRIAL: NCT06929923
Title: An Assessment of Clinical Efficacy of Hypothermic Therapy Following Mild Traumatic Brain Injury (mTBI) in the Adolescent Athlete as Compared to an Untreated Active Control Population
Brief Title: Pro-2-Cool Pivotal Trial II
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA requested changes to study prior to continuation of enrollment
Sponsor: TecTraum Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1380718
Record Dates: First submitted 2025-04-14; First posted 2025-04-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Non-invasive hypothermic therapy
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pro-2-Cool Device (Experimental)
  Interventions: Device: Pro-2-Cool Device
- Standard of Care (No Intervention): "Brain rest"

INTERVENTIONS:
Device: Pro-2-Cool Device — The Pro-2-Cool Device is a non-invasive hypothermic therapy ("cold therapy") device that provides localized cooling of the head and neck. Water and isopropyl alcohol cooled to 6°C by the chiller assembly circulate through the cooling garment to create conductive heat transfer from the scalp and carotid arteries, thus achieving cooling of the brain.
  Arms: Pro-2-Cool Device

SUMMARY:
This study is being conducted to quantify the clinical safety and efficacy of head and neck cooling, using the Pro-2-Cool device, when applied after mTBI injury sustained by adolescents aged 12-21 years, participating in sporting activities.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, non-blinded, dual-arm comparator study enrolling up to a total of 72 patients (approximately 36 patients in the treatment arm and 36 patients in the control arm) following sports-related, mTBI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 12 - 21 years
2. Initial provider visit is within 8 days of mTBI injury
3. Confirmed mTBI diagnosis from sporting activities
4. In generally good health as confirmed by medical history and as determined by site investigator
5. Has a symptom score of at least 7 (analogous of the SCAT5 symptoms score)
6. Has informed consent obtained per protocol and as required per IRB

Exclusion Criteria:

1. Cleared to return to play during initial visit
2. Suffers a serious TBI as evidenced by worsening symptoms, specifically:

   2.1. GCS <14 2.2. Seizure 2.3. Hospitalization 2.4. Existing positive diagnostic testing which include radiology scans that indicate brain bleed 2.5. Slurred speech, which has not resolved within 72 hours of mTBI injury
3. Sustains another head or neck injury at the time of mTBI injury which requires medical treatment
4. History of a serious medical or psychiatric disorder that include:

   4.1. Suicide attempt in the last 6 months 4.2. Unmanaged depression or anxiety 4.3. Hospitalization in the last 6 months for psychiatric treatment
5. History of Reynaud's disease or phenomenon, cold agglutinin disease, cryoglobulinemia, or cryofibrinogenemia
6. Previously diagnosed with a cerebrovascular disorder
7. Is unable to understand the study requirements or the informed consent
8. Currently enrolled in another investigational research study that may confound the results of this study
9. Non-English speaking subjects and parents/legal guardians

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
SCAT-5 change from baseline to the post-72 hour follow-up visit measurement | Baseline to 72-hour follow-up
  Sport Concussion Assessment Tool 5th edition (SCAT-5) is the current standard of practice assessment tool used at the time of injury to diagnose an mTBI.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Reilly, MD, Principal Investigator — Children's Hospital Medical Center of Akron
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Akron Children's Hospital, Akron, Ohio

IPD SHARING:
Plan to Share IPD: No